CLINICAL TRIAL: NCT05672888
Title: Efficacy and Safety of Jaktinib in Patients With COVID-19 Pneumonia.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZGJAK-IIT-002
Record Dates: First submitted 2023-01-04; First posted 2023-01-05 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: COVID-19 Pneumonia
Keywords: Pneumonia; COVID-19 Infection
MeSH Terms: conditions — Pneumonia; COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Jaktinib (Experimental): Jaktinib 100mg BID
  Interventions: Drug: Jaktinib
- Placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Jaktinib — 100mg of Jaktinib (given as two 50mg tablets) administered orally Twice daily(BID) with best available treatment.
  Arms: Jaktinib
Drug: Placebo — Placebo (given as two placebo tablets) administered orally BID with best available treatment.
  Arms: Placebo

SUMMARY:
This was a randomized, double-blind, placebo-controlled parallel study.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age, male or female;
* History of COVID-19 infection within 1 week;
* Subjects with HRCT consistent with viral pneumonia (Judged by investigator) and meeting any of the following criteria: With fever, respiratory symptoms; Shortness of breath present,RR ≥30 breaths/min.
* Clear consciousness, Capable and voluntary informed consent.

Exclusion Criteria:

* Unable to take tablets orally Or suspected hypersensitivity to Jaktinib, drugs of the same class, or their excipients, Patients with severe gastrointestinal dysfunction affecting drug absorption;
* Any person meeting criteria for critical pneumonia;
* Patients considered unsuitable for this trial by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Time to Recovery | Day 1 to Day 28
  Recovery assessed by the National Institute of Allergy and Infectious Diseases Ordinal Scale (NIAID-OS). Time to reach NIAID-OS 1, 2, or 3 for the first time. NIAID-OS: 1 Not hospitalized, no limitations on activities. 2 Not hospitalized, limitation on activities and/or requiring home oxygen. 3 Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care.

SECONDARY OUTCOMES:
Percentage of participants who require invasive mechanical ventilation due to disease progression at Day 3, 7, 1 4 or EOT | Day 3, 7, 14 or EOT
Mortality | Day 1 to Day 28
  Proportion of patients with all-cause mortality at Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Jianya Zhou, Principal Investigator — First Affiliated Hospital of Zhejiang University
Locations (1):
- The First Affiliated Hospital of College of Medicine Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No